CLINICAL TRIAL: NCT06216990
Title: Metastatic or Refractory Soft Tissue Sarcomas and Metronomic Cyclophosphamide: Further Assessment of Efficacy and Safety
Acronym: MeRCY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/704
Record Dates: First submitted 2023-12-14; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Sarcoma; Soft Tissue Sarcoma
Keywords: Cyclophosphamide; Administration, Metronomic
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metronomic Cyclophosphamide's use in monotherapy as a palliative treatment against non-resectable and metastatic Soft Tissue Sarcomas relies on small retrospective cohorts' data.

Current litterature needs external validation of its efficacy and safety profile in these settings of usually frail patients.

The investigators assessed further data and aimed to identify predictive factors of metronomic cyclophosphamide impact in metastatic Soft Tissue Sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18
* with inoperable or metastatic Soft Tissue Sarcoma
* treated with Metronomic Cyclophosphamide
* in 3 cancer care institutions located in 2 French regions (Bourgogne and Franche-Comté)
* between January 2005 and December 2021

Exclusion Criteria:

* patients with bone, chondral sarcomas, desmoid, or gastrointestinal stromal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 with inoperable or metastatic STS, treated with MCP in non curative settings.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of first administration of Metronomic Cyclophosphamide until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-Free Survival is defined as the period from the first day of Metronomic Cyclophosphamide administration until the day of progression or death from any cause Assessment period was from the day of the first day of MCP administration until the first observation of progression or death from any cause.
  Disease progression is defined according to RECIST Ver. 1.1.

SECONDARY OUTCOMES:
Overall Survival | From date of first administration of Metronomic Cyclophosphamide until the date of death from any cause, assessed up to 100 months
  Overall Survival is defined as the period from the first day of Metronomic Cyclophosphamide administration until the day of death from any cause Assessment period was from the day of the first day of Metronomic Cyclophosphamide administration until the first observation of death
Progression Rate | 3 and 6 Months
  Proportions of patients with no reported progression at each time-point (3 and 6 months)
Response Rate (RR) | From date of first administration of Metronomic Cyclophosphamide until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Proportion of Complete Response and Partial Response among the study population from the first day of Metronomic Cyclophosphamide administration until the day of progression or death from any cause.
Control Rate | From date of first administration of Metronomic Cyclophosphamide until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Included Complete Response, Partial Response, and Stable Disease according to RECIST for at least 12 weeks from the first day of Metronomic Cyclophosphamide administration until the day of progression or death from any cause.

OTHER OUTCOMES:
Imputable Toxicity Occurence | From date of first administration of Metronomic Cyclophosphamide until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Occurence, Nature and Grades according to CTCAE 5.0 of clinicians-reported adverse events imputable to metronomic cyclophosphamide

CONTACTS AND LOCATIONS:
Overall Officials: Clément BOLOGNINI, Principal Investigator — CHU Besançon

IPD SHARING:
Plan to Share IPD: Undecided
Clinical data cannot be made publicly available because of privacy issues. However, additional results and aggregated findings are available on reasonable request.